CLINICAL TRIAL: NCT07121426
Title: Effects of Lower Limb Intensive Functional Training on Gait and Balance in Spastic Diplegic Cerebral Palsy Children
Brief Title: Effects of LIFT on Gait and Balance in Spastic Diplegic Cerebral Palsy Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC-UOL-287-01-2023
Record Dates: First submitted 2023-02-18; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2024-02

CONDITIONS: Spastic Diplegic Cerebral Palsy; Gait, Spastic
Keywords: Cerebral palsy, Balance, Gait, Spastic Diplegia
MeSH Terms: conditions — Cerebral Palsy; Gait Disorders, Neurologic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Experimental): Control group will receive Conventional physical therapy and traditional gait training at clinical setting.
  Interventions: Other: Conventional physical therapy
- Intervention Group (Experimental): Experimental group will receive LIFT and conventional physical therapy at home settings provided by their caregivers.
  Interventions: Other: Lower limb Intensive Functional Training; Other: Conventional physical therapy

INTERVENTIONS:
Other: Lower limb Intensive Functional Training — LIFT will help the child in motor learning, skill progression and resistance training to target the strength, proprioception and coordination impairments of the lower extremities. Motor learning will be based on Strength domain (Cycling) . Balance and Coordination domain involves activities such as (ball kicking with alternate legs and Static standing) Proprioception domain (Vertical jumping, sit to stand and cursing) while applying knee-immobilizers if needed.
  Arms: Intervention Group
Other: Conventional physical therapy — Stretching followed by Strengthening program and traditional gait training at clinical setting. Stretching muscles were hip flexors, hip adductors, hamstrings and calf and stretching applied for 30 sec with 30 sec rest for 3-5 times for each muscle group with in pain limit followed by strengthening exercise for week muscle which includes the strengthening of anti-gravity muscles of lower limb they are: Quadriceps, Gluteus maximus and soleus performed in 3 groups. Each group contain 10 rep for each week muscle group.

SUMMARY:
The goal of this Randomized control trial was to evaluate the outcome of limb intensive functional training (LIFT) on gait and balance in spastic diplegic cerebral palsy children with age 3-7 years.

The main questions this study has answered were:

* To access the improvement in children's gait and balance by providing interventions in clinical setting/ standardized environment and then at home environment. This study will check does the improvement in capacity level also improve their performance level in spastic diplegic CP children after getting targeted, activity focused and therapeutic interventions.
* Researcher will compare the effects of intervention on both groups. Control group will receive Conventional physical therapy and traditional gait training at clinical setting while Experimental group will receive LIFT and conventional physical therapy at home settings provided by their caregivers. Both group will receive intervention 5days/week for 20 consecutive weeks.

DETAILED DESCRIPTION:
GMFCS level 3 and MAS level 2 children were eligible to participate in study and Gross Motor Functional Measure (GMFM-88) was used to access Motor Capacity. 10-meter walk test, timed up and go test and 30 sec chair rise tests was used to access Motor Performance.

Method and Procedures of the research were explained to the patients earlier to data collection. Any query was explicated on the spot.

Group A: The Control group received conventional physical therapy (Stretching followed by Strengthening program and traditional gait training) at clinical setting.63 Stretching muscles were hip flexors, hip adductors, hamstrings and calf and stretching applied for 30 sec with 30 sec rest for 3-5 times for each muscle group with in pain limit followed by strengthening exercise for week muscle which includes the strengthening of anti-gravity muscles of lower limb they are: Quadriceps, Gluteus maximus and soleus performed in 3 groups. Each group contain 10 rep for each week muscle group. Conventional Physical therapy applied 5 days/week for consecutive 20 weeks. They were also guided to perform activities at home but they're unbound to do the designed activities freely.

Group B: The experimental group received Lower limb intensive functional training (LIFT) at home environment and conventional physical therapy at clinical setting. LIFT was provided at home environment for 3 hours/day, 5days/week for 5 months.31 A log book was maintained and the goals and strategies were guided to child's parents. 3 hours' treatment was performed in intervals at different time of the day. LIFT helped child in motor learning, skill progression and resistance training to target the strength, proprioception and coordination impairments of the lower extremities.64 Motor learning was based on Strength domain (Cycling) and progression from smooth to rough surface. Balance and Coordination domain involves activities such as (ball kicking with alternate legs and Static standing) and progression was done by increasing accuracy and complexity. Proprioception domain (Vertical jumping, sit to stand and cursing) while knee-immobilizers applied if needed and progression number of repetitions and sets was increased over time. Skill progression was used to challenge the LIFT and make it intensive enough to obtain changes in motor skills and function. AFO's were required during therapy session if needed.

Caregiver were provided proper guidelines before implementing the treatment at home. 3 training sessions was given prior to treatment. A log book was also provided to get the structured record of the treatment. Further videos and mode of tele-rehabilitation was used for supervision and guidance throughout the study. Therapist closely monitored the activities by checking daily logs.

ELIGIBILITY:
Inclusion Criteria:

Children with Spastic diplegic CP with aged 3-7 years Children of both gender Children with MAS level-2 Children with GMFCS level-3 The ability of caregivers to provide one-on-one attention to the child during dailyactivities

Exclusion Criteria:

Visual problems preventing performance of interventions and testing tasks59 Any orthopedic or neuro-surgery done in last 1 year60 Children with any other neurological conditions61 Children with uncontrolled seizures62

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 82 (Actual)
Dates: Start 2023-01-22 (Actual); Primary Completion 2023-06-25 (Actual); Study Completion 2023-07-10 (Actual)

PRIMARY OUTCOMES:
Gross motor function measure | at baseline and after 20 weeks
  GMFM-88 version and clause C, D and E will be used in this study.

SECONDARY OUTCOMES:
10 Meter Walk Test (10mwt) | at baseline and after 20 weeks
  10 MWT accesses performance and used for measurement of walking speed over short duration in meter/sec. It is used to calculate the functional mobility and gait
Timed Up and Go Test (Tug) | at baseline and after 20 weeks
  TUG test evaluates balance, anticipatory postural control, functional mobility and agility in ambulatory children with CP. TUG can be used for differentiation in performance with different types of CP and different levels of GMFCS
30-sec chair rise test | at baseline and after 20 weeks
  The 30-sec chair rise test is used to access leg strength and endurance. 30 sec CRT accessed either by a specific number of sit-ups done in 30 second (e.g.; 10 reps, 5 reps etc.) or total repetitions of sit-ups and down done in 30 sec periods

CONTACTS AND LOCATIONS:
Overall Officials: Umair Ahmed, PhD, Study Chair — University of Lahore
Locations (1):
- Husna Albab, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] 1. Khumlee N, Suriyaamarit D, Boonyong S. Effects of sensory cues on dynamic trunk control in children with spastic diplegic cerebral palsy. Physiotherapy Theory and Practice 2021: 1-8. 2. Ma Y, Liang Y, Kang X, Shao M, Siemelink L, Zhang Y. Gait characteristics of children with spastic cerebral palsy during inclined treadmill walking under a virtual reality environment. Applied bionics and biomechanics 2019; 2019. 3. Zarkou A, Lee SC, Prosser LA, Jeka JJ. Foot and ankle somatosensory deficits affect balance and motor function in children with cerebral palsy. Frontiers in Human Neuroscience 2020; 14: 45. 4. Tatemoto T, Tanaka S, Maeda K, Tanabe S, Kondo K, Yamaguchi T. Skillful cycling training induces cortical plasticity in the lower extremity motor cortex area in healthy persons. Frontiers in Neuroscience 2019; 13: 927.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-01-10): https://cdn.clinicaltrials.gov/large-docs/26/NCT07121426/Prot_SAP_ICF_000.pdf